CLINICAL TRIAL: NCT01714037
Title: A Phase I-II Evaluation of the Safety and Efficacy of the Oral HSP90 Inhibitor Debio 0932 in Combination With Standard of Care in first-and Second-line Therapy of Patients With Stage IIIb or IV Non-small Cell Lung Cancer-the HALO Study (HSP90 Inhibition And Lung Cancer Outcomes)
Brief Title: A Clinical Study on the Safety and Efficacy of Debio 0932 in Combination With Standard of Care in Patients With Non-small Cell Lung Cancer [NSCLC]
Acronym: HALO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0932-201
Record Dates: First submitted 2012-10-03; First posted 2012-10-25 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Safety; Efficacy; HSP90; Debio 0932; Standard of care treatment, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — CUDC 305; Cisplatin; Pemetrexed; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cisplatin, Pemetrexed, Debio 0932 (Experimental): Cisplatin, Pemetrexed, Debio 0932
  Interventions: Drug: Debio 0932; Drug: Cisplatin; Drug: Pemetrexed
- Cisplatin, Gemcitabine, Debio 0932 (Experimental): Cisplatin, Gemcitabine, Debio 0932
  Interventions: Drug: Debio 0932; Drug: Cisplatin; Drug: Gemcitabine
- Docetaxel, Debio 0932 (Experimental): Docetaxel, Debio 0932
  Interventions: Drug: Debio 0932; Drug: Docetaxel

INTERVENTIONS:
Drug: Debio 0932 — Debio 0932 will be administered as daily oral tablets at a starting dose of 250 mg four times per day (QD).
Drug: Cisplatin — Cisplatin 75 mg/m2 body surface area (BSA) will be administered on Day 1 of each 21-day treatment cycle.
  Arms: Cisplatin, Gemcitabine, Debio 0932; Cisplatin, Pemetrexed, Debio 0932
Drug: Pemetrexed — Pemetrexed 500 mg/m2 BSA will be administered on Day 1 of each 21 day treatment cycle.
  Arms: Cisplatin, Pemetrexed, Debio 0932
Drug: Gemcitabine — Gemcitabine 1250 mg/m2 BSA will be administered on Days 1 and 8 of each 21-day treatment cycle.
  Arms: Cisplatin, Gemcitabine, Debio 0932
Drug: Docetaxel — Docetaxel 60 or 75 mg/m2 BSA will be administered on Day 1 of each 21-day treatment cycle.
  Arms: Docetaxel, Debio 0932

SUMMARY:
Part A of this study will investigate the Maximum Tolerated Dose of Debio 0932 in combination with standard of care chemotherapy for the first- and second-line treatment of advanced NSCLC.

DETAILED DESCRIPTION:
Part A of this study will determine the Maximum Tolerated Dose of Debio 0932 in combination with cisplatin/pemetrexed and cisplatin/gemcitabine in treatment-naïve patients with Stage IIIb or IV NSCLC, and with docetaxel in previously treated patients with Stage IIIb or IV NSCLC.

Escalating doses of Debio 0932 will be given to subsequent patients in combination with standard doses of these 3 background chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC with confirmed squamous or non-squamous tumour histology, without known epidermal growth factor receptor (EGFR) mutation
* Advanced or metastatic disease (Stage IIIb or IV)
* Patients to be treated with cisplatin/gemcitabine or cisplatin/pemetrexed: No previous systemic treatment with chemotherapy, targeted therapy or investigational agents (except adjuvant therapy if > 6 months ago); Patients to be treated with docetaxel: ≥ 1 previous treatment with chemotherapy
* Measurable disease by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* ECOG performance score 0-1
* Life expectancy ≥ 3 months
* Adequate bone marrow-, renal- and hepatic function
* LVEF ≥ 55% on cardiac ultrasound

Exclusion Criteria:

* Symptomatic brain metastases
* Gastro-intestinal disorders that could affect drug absorption (including, but not limited to, major abdominal surgery, significant bowel obstruction, ulcerative colitis, Crohn's disease)
* Concurrent treatment with any other systemic anti-cancer therapy
* Serious concomitant uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities | 6 weeks

SECONDARY OUTCOMES:
Change in vital signs and Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Day 1 of each treatment cycle until disease progression or study drug toxicity
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Every treatment cycle until disease progression or study drug toxicity
Incidence of laboratory abnormalities | 2 to 4 times every treatment cycle until disease progression or study drug toxicity
Incidence of treatment discontinuations due to AEs and SAEs | Every treatment cycle until diseases progression or study drug toxicity
Change in left ventricular ejection fraction (LVEF) | Baseline and after 4 weeks of treatment
Pharmacokinetic parameters of Debio 0932 and its metabolite Debio 0932-MET1 | 22 days
Pharmacokinetic parameters of cisplatin/pemetrexed, cisplatin/gemcitabine, and docetaxel | 22 days
Best overall tumor response | 22 days
Pharmacodynamic biomarkers | 22 days
Pharmacogenomic, tumour pharmacogenetic, proteomic, and pharmacogenetic factors predictive of response to Debio 0932 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Isambert, MD, Principal Investigator — Centre GF Leclerc, Dijon, France; Jean-Pierre Delord, PR, Principal Investigator — Institut Claudius Regaud, Toulouse, France; Jèrôme Fayette, MD, Principal Investigator — Centre Léon Bérard, Lyon, France; Jaafar Bennouma, MD, Principal Investigator — Institut de Cancérologie de l'Ouest- Institut René Gauduchau, Nantes, France; Luis Paz-Ares, PR, Principal Investigator — Hospital Universitario Virgen del Rocío, Seville, Spain; Enriqueta Felip, PR, Principal Investigator — Hospital Universitari Vall d'Hebron, Barcelone, Spain; Mariano Provencio, PR, Principal Investigator — Hospital Puerta de Hierro Majadahonda, Madrid, Spain; Ruth Plummer, PR, Principal Investigator — Freeman Hospital, Newcastle, UK
Locations (8):
- France (4):
  - Centre GF Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'Ouest- Institut René Gauduchau, Nantes
  - Institut Claudius Regaud, Toulouse
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Freeman Hospital, Newcastle, United Kingdom

REFERENCES:
- See also: Site Debiopharm SA — http://www.debiopharm.com